CLINICAL TRIAL: NCT06134193
Title: Combination Therapy of HAIC, Surufatinib and Tislelizumab for Unresectable or Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Liang, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230436
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma; Intrahepatic Cholangiocarcinoma; Gallbladder Cancer; Surufatinib; Angiogenesis Inhibitors; Tislelizumab; Antineoplastic Agents, Immunological; Immunotherapy
MeSH Terms: conditions — Carcinoma; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — surufatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC, surufatinib and tislelizumab (Experimental)
  Interventions: Drug: HAIC; Drug: Surufatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: HAIC — hepatic arterial infusion (HAI) of oxaliplatin, fluorouracil, leucovorin (FOLFOX) treatment (Q3W) Oxaliplatin: 85mg/m2 , Day 1 Leucovorin: 200mg/m2, Day 1 Fluorouracil: 400mg/m2, Day1 and 2400mg/m2 continuous arterial perfusion for 46h.
Drug: Surufatinib — 250mg PO d1, Q3W
Drug: Tislelizumab — 200mg IV d1, Q3W

SUMMARY:
This is a single-arm, exploratory study to evaluate the efficacy and safety of HAIC in combination with surufatinib and tislelizumab in the first line treatment of patients with unresectable or metastatic biliary tract cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent should be signed before implementing any trial-related procedures 2. Patients with age ≥18 years ,≤75 years old. 3. ECOG PS scores 0-1 4. Histologically/cytologically confirmed unresectable or metastatic Intrahepatic Cholangiocarcinoma and gallbladder cancer 5. Child Pugh stage A 6. Estimated survival > 12 weeks 7. According to the diagnostic criteria of NCCN(National Comprehensive Cancer Network ) guidelines for intrahepatic cholangiocarcinoma and gallbladder cancer, the patients were diagnosed as intrahepatic cholangiocarcinoma and gallbladder cancer not suitable for radical resection: unable to obtain R0 resection, multiple liver, beyond hilar lymph node metastasis and distant metastasis 8. No systemic therapy for unresectable or metastatic biliary tract cancer; Patients who had received one regimen of adjuvant therapy and had a relapse more than 6 months after the end of chemotherapy were eligible.

  9. At least one measurable lesion according to RECIST V1.1 The diameter of the target lesion was ≥1cm as accurately measured by enhanced magnetic resonance imaging (MRI) or enhanced computed tomography (CT), and the study target lesion had not received previous local treatment (including but not limited to HAIC, radiofrequency ablation, argon-helium knife, radiotherapy, and other local treatment methods) 10. Sufficient organ and bone marrow functions, with the laboratory test values within 14 days before the enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other drugs via intravenous or subcutaneous administrations are allowed for correction treatment within the first 14 days after the laboratory test results are obtained). The specific information is as follows:
  1. Routine blood test: white blood cell ≥ 4.0 × 109/L absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 80 × 109/L; hemoglobin (HGB) ≥ 9.0 g/dL.
  2. Hepatic function: total bilirubin (TBIL) ≤ 3 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN.
  3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or eGFR≥60%,clearance of creatinine (CCr) ≥ 60 mL/min (Cockcroft Gault formula);
  4. Blood coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
  5. Normal cardiac function with left ventricular ejection fraction (LVEF)≥50% measured by two-dimensional echocardiography; 11. Patients were eligible for HAIC surgery as prespecified by the study center, without any contraindications, and could receive HAIC treatment.

  12. Male or female patients of childbearing potential volunteered to use an effective method of contraception, such as dual barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. during the study and for 6 months after the last study medication. "All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnophorectomy, or radioactive ovarian irradiation)."

Exclusion Criteria:

* 1. Participated in other clinical trials of antineoplastic drugs within 4 weeks before enrollment.

  2. History of liver resection, TACE treatment, and any previous immune or targeted therapy; 3. Liver metastases of 70% or more of the total liver volume as determined by the investigator.

  4. History of prior or planned any organ transplantation. 5. Patients with obstructive jaundice who did not reduce jaundice as expected. 6. Other malignant tumors in the past 5 years, excluding basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix.

  7. Patients with confirmed or suspected symptomatic active brain or meningeal metastases.

  8. Received any surgery (except biopsy) or invasive treatment or operation within 4 weeks before enrollment and the surgical incision was not completely healed (except venous catheterization, puncture drainage, etc.).

  9. Electrolyte abnormalities that were judged by the investigator to be clinically significant..

  10. Patients have current drug-uncontrolled hypertension defined as systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg.

  11. Urine routine test showed urinary protein ≥2+, and 24 h urinary protein amount >1.0g.

  12. Patients whose tumors were judged by the investigator to be highly likely to invade vital blood vessels and cause fatal bleeding during the follow-up study.

  13. Patients with evidence or history of significant bleeding tendency within 3 months before enrollment (bleeding within 3 months >30 mL, hematemesis, melena, hematochezia), hemoptysis (within 4 weeks>5 mL of fresh blood); Patients with a history of hereditary or acquired bleeding or coagulopathy. Patients had clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.

  14. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before enrollment; New York Heart Association (NYHA) classification of congestive heart failure >Grade 2; Ventricular arrhythmias requiring medical therapy; Electrocardiogram (ECG) showed QT c interval ≥480 msec.

  15. Women who are pregnant (with a positive pregnancy test before medication) or breastfeeding.

  16. Any other medical condition, clinically significant metabolic abnormality, physical examination abnormality, or laboratory abnormality in which there is reason to suspect that the patient has a disease or condition (e.g., having seizures requiring treatment) that would be inappropriate for use of the study drug, or that would affect interpretation of the study results or place the patient at high risk, in the investigator's judgment.

  17. Severe active or uncontrolled infection (≥CTCAE grade 2 infection), known human immunodeficiency virus (HIV) infection; Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection, i.e., HBV DNA positive (> 1×104 copies /mL or >2000 IU/ mL), known hepatitis C virus (HCV) infection with positive HCV RNA (>1×103 copies /mL), or other hepatitis, cirrhosis.

  18. Patients with any active, known or suspected autoimmune disease (including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, hypophysitis, hyperthyroidism, etc.) Patients with any active, known or suspected autoimmune disease (including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, hypophysitis, hyperthyroidism, etc).

  19. Known allergic reactions to other monoclonal antibodies or to any component of surufatinib.

  20. According to the investigator's judgment, patients have other factors that may affect the results of the study or lead to the forced termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment, family or social factors, etc., which will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) per RECIST v1.1 | From baseline to primary completion date, about 18 months
  Defined as a duration from the date of initial treatment to disease progression or death of any cause

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 3 months
  Defined as the sum of the complete response and partial response rate
Disease control rate (DCR) per RECIST v1.1 and mRECIST | From baseline to primary completion date, about 3 months
  Defined as the sum of the complete response, partial response and stable disease
Overall survival (OS) | From baseline to primary completion date, about 24 months
  Defined as a duration from the date of initial treatment to death of any cause
Conversion to surgical resection rate | From baseline to primary completion date, about 6 months
  Defined as the proportion of patients who were successfully converted to radical resection with negative hepatic margins after the study treatment regimen was calculated
Incidence rate of adverse events | From baseline to primary completion date, about 18 months
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No